CLINICAL TRIAL: NCT04936477
Title: Functional Morphometry and Ventilation Perfusion Ratio to Estimate the Alveolar Surface Area in Prematurely Born Infants
Brief Title: Ventilation-perfusion (V/Q) Ratio and Alveolar Surface Area in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KCH20-138
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-08

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment of alveolar surface area by functional morphometry (Experimental): Non-invasive measurements of V/Q
  Interventions: Other: Calculation of ventilation-perfusion ratio

INTERVENTIONS:
Other: Calculation of ventilation-perfusion ratio — Three to five paired measurements of fraction of inspired oxygen and peripheral oxygen saturations.
  Insertion of mainstream capnograph with combined pressure and flow sensor to perform end-tidal capnography measurement.
  Echocardiogram to assess intra-cardiac shunting.

SUMMARY:
To non-invasively estimate the alveolar surface area of the lungs of prematurely born infants by taking measurements of oxygen and carbon dioxide and utilizing functional morphometry.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Congenital or chromosomal anomalies

Ages: 22 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Calculation of the alveolar surface area in prematurely born infants using validated functional morphometry | One year

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided